CLINICAL TRIAL: NCT03855956
Title: A Randomized, Double-blind, Controlled, Clinical Food Study to Evaluate the Effect of KB174 Compared to an Easily Digestible Polysaccharide on Function and Structure of the Gut Microbiome in Subjects With Well-compensated Cirrhosis
Brief Title: Clinical Food Study to Evaluate the Effect of KB174 on the Gut Microbiome in Subjects With Well-compensated Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: K022-118
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Early Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KB174 Arm (Experimental): KB174 is a novel mixture of oligosaccharides.
  Interventions: Other: KB174
- Maltodextrin Arm (Other): Maltodextrin is a commercially available easily digestible polysaccharide.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: KB174 — KB174 is a novel mixture of oligosaccharides.
  Arms: KB174 Arm
Other: Maltodextrin — Maltodextrin is a commercially available easily digestible polysaccharide.
  Arms: Maltodextrin Arm

SUMMARY:
This randomized, double-blind, controlled, clinical food study aims to explore KB174, a novel mixture of oligosaccharides, and maltodextrin, an easily digestible polysaccharide, on gut microbiome structure and function in subjects with well-compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent
* Be male or female, 18 to 70 years of age (inclusive)
* Have a body mass index (BMI) ≥ 20.0 and < 40.0 kg/m2
* Well-compensated cirrhosis
* Negative for hepatocellular carcinoma (HCC)
* Adequate safety laboratory values at Screening.
* Be willing to maintain a stable diet throughout the course of the study, and willing to continue usual exercise routine
* If of child bearing potential must follow contraceptive requirements of the protocol
* Have reliable internet access

Exclusion Criteria:

* Have evidence of decompensated liver disease.
* History or active GI disease.
* Prior solid organ transplantation, including liver transplantation or on liver transplant waiting list.
* Subject has a history of drug and/or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in 15N in urine in response to an amino acid challenge, from Baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 28.
  Change in 15N in urine in response to an amino acid challenge during Baseline (pre-study compound consumption) versus post-28-day study compound compound consumption.

SECONDARY OUTCOMES:
Change in 15N in stool in response to an amino acid challenge, from Baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in 15N in stool in response to an amino acid challenge during Baseline (pre-study compound consumption) versus post 28-day study compound consumption.
Change in total nitrogen in blood in response to an amino acid challenge, from Baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 27.
  Change in total nitrogen in blood in response to an amino acid challenge during Baseline [pre-study compound consumption] versus post 28-day study compound consumption.
Change in total nitrogen in urine in response to an amino acid challenge, from Baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in total nitrogen in urine in response to an amino acid challenge during Baseline [pre study compound consumption] versus post 28-day study compound consumption.
. Change in total nitrogen in stool in response to an amino acid challenge, from Baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in total nitrogen in stool in response to an amino acid challenge during Baseline [pre study compound consumption] versus post 28-day study compound consumption.
Change in ammonia in blood for KB174 compared to Maltodextrin. | Day -3 to Day 43.
  Change in ammonia in blood from Baseline to end of study for KB174 compared to maltodextrin
Change in total urea in urine in response to an amino acid challenge from baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in total urea in urine in response to an amino acid challenge during baseline [pre study compound consumption] versus post 28-day compound consumption.
Change in 15N-urea in urine in response to an amino acid challenge from baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in 15N-urea in urine in response to an amino acid challenge from baseline [pre study compound consumption ] versus post 28-day compound consumption.
Change in 15N-urea in stool in response to an amino acid challenge from baseline to Tracer Period 2, for KB174 compared to maltodextrin. | Day -3 to Day 29.
  Change in 15N-urea in stool in response to an amino acid challenge from baseline [pre study compound consumption ] versus post 28-day compound consumption.
Incidence of treatment-emergent adverse events from baseline to end of study. | Day -7 through Day 43 visit.
Incidence of serious adverse events from base baseline to end of study. | Day -7 through Day 43.
Change in Gastrointestinal Tolerability Questionnaire (GITQ) through the collection of daily patient questionnaires. | Day -7 through Day 43.
  Evaluate the effect of KB195 on self-report questionnaires including the Gastrointestinal Tolerability Questionnaire, an assessment of the frequency and severity of GI symptoms, e.g., gas, abdominal pain, calculated on a scale from 0 (None/Not applicable) to a maximum score of 60 (Severe/Much more than usual) for all questions.
Change in Bristol Stool Scale (BSS) through the collection of daily patient questionnaires | Day -7 through Day 43.
  Evaluate the effect of KB195 on self-report questionnaires including the Bristol Stool Scale, an assessment of stool consistency on a scale from 1 (separate hard lumps, like nuts, hard to pass) through 7 (watery, no solid pieces, entirely liquid).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Centers of America, Hollywood, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Marquez Clinical Site Partners, LLC Florida Premier Research Institute, Winter Park, Florida
  - Delta Research Partners, Monroe, Louisiana

IPD SHARING:
Plan to Share IPD: No